CLINICAL TRIAL: NCT05570513
Title: Relation of IL23R and IL17A Gene Polymorphisms Plus Serum Levels of IL23 and IL17A to Rheumatoid Arthritis Susceptibility and Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Salah Mohamed Hussein, Assistant lecturer at Medical Microbiology and Immunology Faculty of Medicine, Assiut university, Assiut University
Other Study IDs: IL23 and IL17A in RA
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assess the impact of rs2201841 and rs2275913 single nucleotide polymorphism of host genes IL-23R and IL-17A respectively on susceptibility of rheumatoid arthritis .

Determine serum levels of IL-23 and IL-17A using ELISA test to investigate their correlation to rheumatoid arthritis disease activity .

Compare the 4 biomarkers IL-23R and IL-17A genetic polymorphism and levels of IL-23 and IL-17A as predictors of rheumatoid arthritis susceptibility and disease activity .

DETAILED DESCRIPTION:
Rheumatoid arthritis an autoimmune disease that is associated with progressive disability, systemic complications and socioeconomic costs. RA affects 0.5-1% of the human population making it one of the most common autoimmune disorders. The incidence of RA increases with age, affecting about 6% of the population over 65 years old. Women are more affected than men in a ratio of 3:1 (1) .

The synovitis in RA is characterized by massive cellular infiltration of the synovium consisting mainly of leukocytes such as T and B cells, macrophages, granulocytes and dendritic cells, together with the increased local production of proinflammatory cytokines and chemokines, eventually leading to the destruction of the joint and bone (2) .

Th-17 starts producing IL-17 and IL-22 which in turn stimulate fibroblast-like synoviocytes (FLS) to secrete IL-8, IL-6, CCL20 and CXCL8 causing inflammation, while the macrophages secreted TNF-α results in IL-23 production from FLS, forming a positive feedback loop that maintains the production of IL-17 and IL-22 from Th-17 (3) . Both IL-17 and IL-22 are able to induce osteoclast differentiation from osteoclast progenitor either directly, or by elevating Receptor activator of nuclear factor kappa-B ligand (RANKL) on CD4+ and Th-17 which upon ligation with the RANK receptor on osteoclast progenitor stimulates osteoclast differentiation. Osteoclasts are a main cause of bone erosion (4).

However, advances in understanding the pathogenesis of the disease have fostered the development of new therapeutics, with improved outcomes (5) . Overall, current treatment strategies for RA tend to involve targeting pro-inflammatory cytokines, and thereby the activation process of inflammation, rather than functioning to boost pathways that orchestrate the suppression and resolution of inflammation (6) .

IL-23 is a pro-inflammatory cytokine that belongs to the IL-12 family, together with IL-12, IL-27, IL-35, and IL-39 (7) .Its actions are mainly mediated by the CD4 T helper subset Th17, a distinct subpopulation of gamma/delta T cells (Tγδ17 cells), subsets of natural killer T (NKT) cells, and type 3 innate lymphoid cells (ILC3s) (8) The main role of IL-23 is to induce the differentiation of αβ T CD4+ naïve cells (Th0 cells) in T helper type 17 (Th17 cells), (9) which are considered pivotal players in autoimmunity (10) . The IL-23 receptor (IL-23R) is a heterodimeric receptor composed of 2 subunits: IL-12Rβ1, in common with the IL-12 receptor (IL-12R) and IL-23Rα, specific to IL-23 signaling (11). The Th17 subset of T-helper cells is pro-inflammatory, plays vital roles in host defense and is involved in the pathogenesis of RA primarily by secreting IL-17 (12) .

SNP is a single base pair mutation at a specific locus, usually consisting of two alleles (where the rare allele frequency is > 1%). The genetic factors account for 50-60% of all RA cases (13) . Some researchers have reported the relationship between IL-23R gene polymorphisms and RA risk but got no consistent results . Therefore, this study will search the role of IL-23R gene rs11209026 polymorphisms in individual susceptibility to RA . Many different genetic variants with functional gene polymorphisms may play a culprit role in the underlying pathogenetic mechanisms (14) .

IL-23R gene variants increase susceptibilities to autoimmune disease in patients with psoriasis, inflammatory bowel disease, and multiple sclerosis (15) . IL-17A is a promising target for anti-cytokine therapy in autoimmune arthritis (16).

In recent years, the associations between IL-17A polymorphisms and RA risk have been studied in various populations by many researchers, (17) with the most frequent variant being IL-17A rs2275913 .

The IL-17A rs2275913 polymorphism is located in the promoter region of the IL-17A gene, and cells with the 197A positive allele (genotypes GA/AA) secreted more IL-17A than cells with the 197A negative allele (18) .

Hence, the IL-17A rs2275913 polymorphism results in more efficient secretion of IL-17A, which may be a potential mechanism by which this polymorphism can increase the risk of developing RA. Many studies hypothesized that rs2201841 and rs2275913 SNP of IL-23R and IL-17A genes respectively have good prediction role for RA susceptibility and severity . Genetic and experimental data support the concept that the activation of IL-23/IL-17 axis contributes to the development of a series of inflammatory rheumatic diseases, including, rheumatoid arthritis (RA). It rapidly became a critical target of research to determine predictors of severity to guide therapeutic intervention .

ELIGIBILITY:
Inclusion Criteria:

* A total of 45 Patients fulfilling the 2010 Classification Criteria of the American college of Rheumatology/European League against Rheumatism (ACR / EULAR) will be included in the study.

The patients will be recruited from department of Physical medicine, Rheumatology & Rehabilitation, Assiut University Hospital.

Exclusion Criteria:

* Patients with other connective tissue diseases (e.g. SLE, systemic sclerosis (SS), BD,...etc), associated autoimmune diseases, chronic liver or kidney diseases, or genetic diseases will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 90 subjects (45 rheumatoid arthritis patients and 45 healthy control)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-04 (Estimated); Primary Completion 2025-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
serum levels of IL23 and IL17A and its Relation to Rheumatoid Arthritis susceptibility and activity | 3 years